CLINICAL TRIAL: NCT00364039
Title: A Phase 1 Double-Blind, Placebo-Controlled Single Center Trial to Assess the Safety, Tolerability and Pharmacokinetics of Single Dose and Multiple Dose Escalations of AV650 in Healthy Subjects
Brief Title: Study to Examine the Safety, Tolerability, and Pharmacokinetics of AV650
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avigen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: AV650-012
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Last update posted 2007-02-28 (Estimated); Status verified 2007-02

CONDITIONS: Healthy Subjects

INTERVENTIONS:
Drug: AV650

SUMMARY:
The purpose of this study is to determine the safety and tolerability of AV650 in healthy subjects given single and multi-doses under fasted and fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking
* Body mass index between 18.5 and 29.9 kg/m2 or body mass index greater than 29.9 kg/m2 with good to excellent body fat percentage

Exclusion Criteria:

* Known hypersensitivity to lidocaine or non-steroidal anti-inflammatory agents (NSAIDS)
* History of clinically significant cardiovascular, pulmonary, endocrine, neurological, metabolic, or psychiatric disease
* History of HIV or Hepatitis B
* History of symptomatic hypotension
* History of mental illness, drug addiction, drug abuse or alcoholism
* History of cancer
* History of inflammatory arthritis (rheumatoid, lupus, psoriatic arthritis)
* Current use of immunosuppressive therapy (systemic steroids, cyclosporine) or use of nasal or topical steroids
* History of gastric or duodenal ulcer disease
* History of severe physical injury, direct impact trauma or neurological trauma within 6 months of Study Day 1
* Female subjects who are pregnant or nursing
* Have donated blood within 90 days of Study Day -1
* Have received an investigational drug within 90 days of Screening
* Require regular use of antihistamines, H2 blockers (such as cimetidine, ranitidine), TCAs or SSRIs or who have taken these medications witin 14 days of Study Day 1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-08

PRIMARY OUTCOMES:
Safety
Tolerability

SECONDARY OUTCOMES:
Pharmacokinetic profile
Sedation and reaction time changes

CONTACTS AND LOCATIONS:
Overall Officials: Stephan A. Bart, M.D., Principal Investigator — SNBL Clinical Pharmacology Center
Locations (1):
- SNBL Clinical Pharmacology Center, Baltimore, Maryland, United States